CLINICAL TRIAL: NCT05967156
Title: Safety and Efficacy of Empagliflozin on Heart Failure Dialysis Patients
Brief Title: Empagliflozin in Heart Failure Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Assistant Professor, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBMU--
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Hemodialysis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empagliflozin (Experimental): Heart failure dialysis patients will be treated with Empagliflozin
  Interventions: Drug: Empagliflozin10Mg Tab

INTERVENTIONS:
Drug: Empagliflozin10Mg Tab — 10 mg daily
  Other Names: Abide

SUMMARY:
Empagliflozin is not still approved for glomerular filtration rate < 20 cc/min/1.73m2. Considering the cardiac and renal benefits of this drug, the evaluation of the safety and efficacy of Empagliflozin for heart failure dialysis patients seems to be mandatory.

DETAILED DESCRIPTION:
Heart failure dialysis patients with residual renal function will be followed up on Empagliflozin based on echocardiographic parameters, pro-brain natriuretic peptide levels, diuresis volume, and serum acidity.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure on dialysis with residual renal function

Exclusion Criteria:

* Dialysis patients with no residual urine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Brain Natriuretic Peptide | one month after administration
  serum level

CONTACTS AND LOCATIONS:
Overall Officials: Dalili, Principal Investigator — SMBU
Locations (1):
- Nooshin Dalili, Tehran, Iran